CLINICAL TRIAL: NCT00046683
Title: A Phase III Study to Evaluate the Efficacy and Safety of Front-Line Therapy With Alemtuzumab (Campath, MabCampath) vs Chlorambucil in Patients With Progressive B-Cell Chronic Lymphocytic Leukemia
Brief Title: Efficacy/Safety of Frontline Alemtuzumab (Campath, MabCampath) vs Chlorambucil in Patients With Progressive B-Cell Lymphocytic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAM307
Record Dates: First submitted 2002-10-01; First posted 2002-10-02 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: B Cell Chronic Lymphocytic Leukemia
Keywords: Adult acute leukemia; Adult chronic leukemia; Childhood leukemia; Campath; Alemtuzumab
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Alemtuzumab

INTERVENTIONS:
Drug: alemtuzumab

SUMMARY:
This is a Phase III, open-label, multicenter, randomized, comparative study of Campath versus chlorambucil as front line therapy in patients with progressive B-Cell Lymphocytic Leukemia (B-CLL). Eligible patients must have previously untreated, Rai stage I-IV disease, and be experiencing progression of their B-CLL requiring treatment. Patients who meet all eligibility criteria may be randomized on a 1:1 basis to receive either Campath or chlorambucil. An estimated 284 patients (142 per treatment arm) from approximately 40 or more investigational sites will be randomized to one of the two treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed diagnosis of B-CLL with CD5, CD19, or CD23 positive clone.
* Rai Stage I through IV disease with evidence of progression as evidenced by the presence of one or more of the following:1. Disease-related B symptoms (fever of greater than 38 celsius (100.5 F) for greater than or equal to 2 weeks without evidence of infection, night sweats without evidence of infection, weight loss >10% within previous 6 months. 2. Evidence of progression marrow failure as manifested by: a. decrease in hemoglobin to <11g/dL or b. decrease in platelet count to <100x10 to the ninth/L within the previous 6 months or c. decrease in absolute neutrophil count (ANC) to <1.0x10 to the ninth/L within the previous 6 months. 3. Progressive splenomegaly to >2 cm below the left costal margin or other organomegaly with progressive increase over 2 consecutive clinic visits greater than or equal to 2 weeks apart. 4. Progressive lymphadenopathy with at least 5 sites of involvement with either two nodes at least 2cm in longest diameter or one node greater than or equal to 5cm in longest diameter with progressive increase over 2 consecutive visits greater than or equal to weeks apart. 5. Progressive lymphocytes with an increase of >50% over a 2-month period, or an anticipated doubling time of less than 6 months.
* Received no previous chemotherapy for B-CLL.
* Life expectancy of at least 12 weeks.
* WHO performance status of 0, 1, or 2.
* Serum creatinine less or equal to 2.0 times the institutional upper limit of normal (ULN) value.
* Adequate liver function as indicated by a total bilirubin, AST, and ALT less or equal to 2 times the institutional ULN value, unless directly attributable to the disease.
* Female patients with childbearing potential must have a negative serum pregnancy test within 2 weeks prior to randomization. Male and female patients must agree to use an effective contraceptive method while on study treatment, if appropriate, and for a minimum of 6 months after study therapy.
* Signed, written informed consent.
* 18 years of age or older.

Exclusion Criteria:

* ANC less than 500 million per liter or platelet count less than 10 billion per liter.
* Medical condition requiring chronic use of oral corticosteroids.
* Autoimmune thrombocytopenia.
* Previous bone marrow transplant.
* Use of investigational agents within previous 30 days.
* Positive for HIV.
* Past history of anaphylaxis following exposure to rat or mouse-derived complementary determining region (CDR) grafted humanized monoclonal antibodies.
* Active infection.
* Serious cardiac or pulmonary disease that could interfere with their ability to participate in the study.
* Recent documented (with in 2 years) of active tuberculosis (TB), current active TB, or currently receiving anti-tuberculosis medication.
* Active secondary malignancy.
* Central nervous system involvement with CLL.
* Positive quantitative CMV by PCR assay (using the laboratory normal ranges).
* A diagnosis of mantle cell lymphoma.
* Other severe, concurrent diseases or mental disorders.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284
Dates: Start 2001-07; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Campath vs. chlorambucil

SECONDARY OUTCOMES:
survival comparison

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (20):
- United States (20):
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Fort Myers, Florida
  - Tampa, Florida
  - Hines, Illinois
  - Louisville, Kentucky
  - Paducah, Kentucky
  - Lafayette, Louisiana
  - Jackson, Mississippi
  - Tupelo, Mississippi
  - Jefferson City, Missouri
  - Kansas City, Missouri
  - Billings, Montana
  - Omaha, Nebraska
  - New Hyde Park, New York
  - Rochester, New York
  - Durham, North Carolina
  - Sioux Falls, South Dakota
  - San Antonio, Texas
  - Norfolk, Virginia

REFERENCES:
- See also: Related Info — http://www.genzyme.com